CLINICAL TRIAL: NCT06759519
Title: An Observational Multicenter Retrospective-prospective Study of Patients With Active Moderate to Severe SLE
Brief Title: Clinical and Demographic Features of Patients With Moderate to Severe Active Systemic Lupus Erythematosus in Russia
Acronym: SEVERUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00092
Record Dates: First submitted 2024-08-28; First posted 2025-01-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic lupus erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multicenter observational retrospective-prospective study consisting of retrospective and prospective phases. Trial will include 2 visits for obtaining the patient's demographic and clinical data: the 1st is retrospective and the 2nd is prospective. The study will involve approximately 50 sites of the Russian Federation; in each site about 20 patients will be recruited. The total planned size of study population will be approximately 1000 patients enrolled to the retrospective phase of the study, from which ~ 600 patients will be enrolled to the prospective phase.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic autoimmune rheumatic disease with variable clinical manifestations and an unpredictable course, affecting any organs or systems, which quite often develops over several months or years, with persistent or, conversely, rapidly changing clinical manifestations, an undulating course, alternating remissions and flares.

Currently, in Russia there is no exact data on the number of patients with active moderate to severe SLE in the population, since there is no unified system for regular monitoring of patients with SLE in the country. The systematic information about complications and comorbidities, about the treatment approaches and their effectiveness in the Russian population is also absent.

The Russian Federation consists of 85 regions with a total population of more than 145 million people. The regions differ in ethnic composition, age, gender, climate, ecology, economic level, prevalence of SLE in general and moderate to severe SLE in particular.

Thus, there is a need to perform a large-scale observational study in regions of the country with a sufficient size of population to obtain information on moderate to severe SLE epidemiology, clinical and demographic characteristics, to describe main clinical outcomes and evaluate existing associations between observed treatment patterns and clinical outcomes in real clinical practice.

Trial will include 2 visits for obtaining the patient's demographic and clinical data: the 1st is retrospective and the 2nd is prospective. To allow wide data coverage the study will involve approximately 50 sites of Russian Federation; in each site about 20 patients will be recruited.

Overall expected duration of the study (from the first patient inclusion to the last patient last visit) is about 13 months or until 1000 patients will be included in the retrospective phase and ~ 600 patients - in the prospective phase This observational study does not imply any intervention into a routine clinical practice, including choice of treatment modality or special methods of investigation.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the retrospective phase are:

1. Patients with the diagnosis of SLE (ICD code: M32) confirmed by medical records;
2. Patients with availability of data of at least one visit to the clinic in the medical records in the last 24 months prior to inclusion;
3. Age ≥ 18 years at the time of last patient's visit to the clinic.

   Additional inclusion criteria for the prospective phase are:
4. Signed and dated written informed consent in accordance with ICH-GCP and local law prior to inclusion in the prospective phase of the study;
5. Disease activity measured with SLEDAI-2K ≥ 6 despite of standard treatment at the time of inclusion in the prospective phase of the study

Exclusion Criteria:

Exclusion criteria for the retrospective phase are:

1. Regular use of genetically engineered biological drugs for SLE treatment within the last 24 months prior to inclusion;
2. Participation in any interventional trial since the last patient's visit to the clinic;
3. Presence of lupus nephritis class III/IV ± V at the moment of the last patient's visit to the clinic;
4. Presence of neuropsychiatric lupus at the moment of the last patient's visit to the clinic.

   Additional exclusion criteria for the prospective phase are:
5. Current use of genetically engineered biological drugs for SLE treatment;
6. Current participation in any interventional trial;
7. Presence of lupus nephritis Class III/IV ± V at the moment of patient's visit;
8. Presence of neuropsychiatric lupus at the moment of patient's visit;
9. An acute or chronic disease that, in the opinion of the investigator, limits the ability of patient to provide data on his/her health or participate in this study or influence the interpretation of the results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is planned to enrol ~ 600 patients with moderate to severe SLE. Before that approximately 1000 patients with confirmed diagnosis of SLE will be screened (retrospective phase).
Sampling Method: Probability Sample
Enrollment: 621 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
disease activity status at the time of patient visit to the doctor measured with SLEDAI-2K, expressed as the mean SLEDAI-2K total score at Visit 2. | patient's visit to the doctor (Visit 2 -prospective data collection)
  In order to achieve primary objective, the mean SLEDAI-2K total score at Visit 2 will be calculated among patients with moderate to severe SLE (i.e. SLEDAI-2K total score ≥6 measured on the Visit 2) who provided informed consent and were enrolled to the prospective phase. The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a clinical index for the measurement of disease activity in SLE. The modified index SLEDAI-2K was introduced and validated in 2002; it allows the documentation of persistent activity disease in rash, mucous membrane ulcers, alopecia, and proteinuria. 4 activity categories have been defined on the basis of the SLEDAI-2K total score (higher scores indicate more damage): no activity (0 points); low activity (1-4 points); moderate activity (5-10 points), and high activity (>10 points).

SECONDARY OUTCOMES:
1. Mean age at the inclusion into the study | inclusion into the study
2. Proportion of patients aged 18-44, 45-64, and ≥65 years at the inclusion into the study | inclusion into the study
3. Mean age at the SLE diagnosis | within 24 months prior to inclusion into the study
4. Mean and median SLE duration, years | from the SLE diagnosis to the Visit 1
5. Proportion of men and women | inclusion of a patient into retrospective part of the study (Visit 1)
6. Proportion of patients from each residential region of Russia | inclusion of a patient into retrospective part of the study (Visit 1)
7. Mean SLEDAI-2K activity total score at Visit 1 (if available) | inclusion of a patient into retrospective part of the study (Visit 1)
  The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a clinical index for the measurement of disease activity in SLE. The modified index SLEDAI-2K was introduced and validated in 2002; it allows the documentation of persistent activity disease in rash, mucous membrane ulcers, alopecia, and proteinuria. 4 activity categories have been defined on the basis of the SLEDAI-2K total score (higher scores indicate more damage): no activity (0 points); low activity (1-4 points); moderate activity (5-10 points), and high activity (>10 points).
8. The proportion of patients with each SLE activity category based on SLEDAI-2K total score at Visit 1 (if available): | inclusion of a patient into retrospective part of the study (Visit 1)
  * No activity (total score 0);
  * Low (total score 1-4);
  * Moderate (total score 5-10);
  * High (total score >10); The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a clinical index for the measurement of disease activity in SLE. The modified index SLEDAI-2K was introduced and validated in 2002; it allows the documentation of persistent activity disease in rash, mucous membrane ulcers, alopecia, and proteinuria. 4 activity categories have been defined on the basis of the SLEDAI-2K total score (higher scores indicate more damage): no activity (0 points); low activity (1-4 points); moderate activity (5-10 points), and high activity (>10 points).
9. The proportion of patients with each SLE activity category based on SLEDAI-2K total score at Visit 2: | patient's visit to the doctor (prospective part of the study)
  * Moderate (total score 5-10);
  * High (total score >10). The Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) is a clinical index for the measurement of disease activity in SLE. The modified index SLEDAI-2K was introduced and validated in 2002; it allows the documentation of persistent activity disease in rash, mucous membrane ulcers, alopecia, and proteinuria. 4 activity categories have been defined on the basis of the SLEDAI-2K total score (higher scores indicate more damage): no activity (0 points); low activity (1-4 points); moderate activity (5-10 points), and high activity (>10 points).
10. Mean SLICC/ACR damage index score by each domain and total score at Visit 2 | patient's visit to the doctor (Visit 2 -prospective data collection)
  The Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR damage index or SDI) is a 42-item questionnaire concerning long-term damage due to SLE in 12 organ systems for use in clinical research studies [14, 15]. The global score (range from 0 to 49, with higher scores indicating more damage) is the sum of the scores for all 12 organ systems.
11. The proportion of patients with various organ domain involvement: | Retrospective and prospective data collection (Visit 1, Visit 2)
  1. Skin and mucosa involvement;
  2. Joints involvement;
  3. Hematological disorders;
  4. Immunological activity;
  5. Renal involvement;
  6. Serositis (pleurisy, pericarditis etc.).
12. The proportion of patients with various comorbidities and concomitant treatment | patient's visit to the doctor (Visit 2 -prospective data collection)
13. The proportion of patients with various groups of SLE treatment medications in anamnesis (at Visit 1) | inclusion of a patient into retrospective part of the study (Visit 1)
14. The proportion of patients taking various groups and drugs of SLE treatment medications (at Visit 2); | patient's visit to the doctor (Visit 2 -prospective data collection)
15. The mean (median) of oral glucocorticosteroids (OGCS) daily dose, | Retrospective and prospective data collection (Visit 1, Visit 2)
  mg/day (prednisolone equivalent) (evaluated in patients who are taking OGCS);
16. The proportion of patients received OGCS daily dose (prednisolone equivalent) more than 5 mg/day; | Retrospective and prospective data collection (Visit 1, Visit 2)
17. Proportion of patient receiving immunosuppressive agents (azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil, cyclosporine, calcineurin inhibitors etc.) as a single agent or combination | Retrospective and prospective data collection (Visit 1, Visit 2)
18. The mean value of immunological laboratory parameters | Visit 2 (within around a year from inclusion into the study)
  C3, C4, anti-dsDNA, ANA
19. The mean value of hematology laboratory parameters | patient's visit to the doctor (Visit 2 -prospective data collection)
  leukocytes, platelets
20. The proportion of patients with leukopenia <4,000/mm³; | patient's visit to the doctor (Visit 2 -prospective data collection)
21. The proportion of patients with thrombocytopenia <100,000/mm³. | patient's visit to the doctor (Visit 2 -prospective data collection)

CONTACTS AND LOCATIONS:
Locations (32):
- Russia (32):
  - Research Site, Barnaul
  - Research Site, Belgorod
  - Research Site, Chelyabinsk
  - Research Site, Grozny
  - Research Site, Irkutsk
  - Research Site, Izhevsk
  - Research Site, Kaliningrad
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnodar
  - Research Site, Makhachkala
  - Research Site, Moscow
  - Research Site, Murmansk
  - Research Site, Nizny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Orenburg
  - Research Site, Penza
  - Research Site, Perm
  - Research Site, Petrozavodsk
  - Research Site, Ryazan
  - Research Site, Saint-Petrburg
  - Research Site, Samara
  - Research Site, Saransk
  - Research Site, Saratov
  - Research Site, Surgut
  - Research Site, Tula
  - Research Site, Ufa
  - Research Site, Ulyanovsk
  - Research Site, Volgograd
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org